CLINICAL TRIAL: NCT02159196
Title: Effectiveness of Routine Nebulization of Mucolytics and Bronchodilators in Mechanically Ventilated Intensive Care Patients'
Brief Title: Effectiveness of Routine Nebulization of Mucolytics and Bronchodilators During Mechanical Ventilation
Acronym: Nebulae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr. Marcus J. Schultz, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nebulae
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; nebulisation; respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Acetylcysteine; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetylcysteine and salbutamol (Active Comparator): Nebulisation of 3 mL-solution of acetylcysteine (fluimucil 100mg/ml, a mucolytic) and a 2.5 mL solution containing salbutamol (ventolin 2.5 Nebules 2.5mg/2.5 ml, a bronchodilator), administered every 6 hours (i.e., 4 times per day) within 24 hours after initiation of ventilation until tracheal extubation.
  Interventions: Drug: acetylcysteine and salbutamol
- acetylcysteine or salbutamol (Experimental): Nebulisation on strict clinical indications; nebulisation of 3 mL-solution of acetylcysteine (fluimucil 100mg/ml, a mucolytic) in case of occurrence of persistent thick and tenacious sputum and only after active humidification is set.
  Nebulisation of 2.5 mL solution containing salbutamol (ventolin 2.5 Nebules 2.5mg/2.5 ml, a bronchodilator) in case of occurrence of bronchospasm.
  Interventions: Drug: acetylcysteine; Drug: salbutamol

INTERVENTIONS:
Drug: acetylcysteine and salbutamol — routine nebulisation of a 3 mL-solution of acetylcysteine (fluimucil 100mg/ml) and a 2.5 mL solution containing salbutamol (ventolin 2.5 Nebules 2.5mg/2.5 ml) four times daily
  Other Names: 3 mL fluimucil 100mg/ml; 2.5 mL ventolin 2.5 Nebules 2.5mg/2.5 ml
  Arms: acetylcysteine and salbutamol
Drug: acetylcysteine — nebulisation of acetylcysteine on strict clinical indications only', i.e. in case of occurrence of persistent thick and tenacious sputum
  Other Names: 3 mL-solution of acetylcysteine (fluimucil 100mg/ml)
  Arms: acetylcysteine or salbutamol
Drug: salbutamol — nebulisation of salbutamol on strict clinical indications only', i.e. in case of occurrence of bronchospasm
  Other Names: 2.5 mL salbutamol (ventolin 2.5 Nebules 2.5mg/2.5 ml
  Arms: acetylcysteine or salbutamol

SUMMARY:
The purpose of this multi-center randomized controlled non-inferiority trial is to determine the effect of a strategy using routine nebulisation of mucolytics and bronchodilators (four times daily) as compared to a strategy using nebulisation of mucolytics or bronchodilators only on clinical indication (i.e. occurrence of persistent thick and tenacious sputum or bronchospasm) in mechanically ventilated intensive care patients. The investigators will examine the effects in terms of ventilator-free days, defined as the number of days alive and free of ventilation at day 28 after start of ventilation.

We hypothesize that a strategy that uses nebulisation of mucolytics or bronchodilators only on clinical indication not to be inferior to a strategy using preventive nebulisation of mucolytics or bronchodilators with regard to the number of ventilator free days in ICU patients at day 28.

DETAILED DESCRIPTION:
Detailed Description clinical trials.gov:

Design: This will be an investigator-initiated, multi-center, randomized, controlled, parallel two group, non-inferiority trial in intubated and ventilated adult ICU patients. A total of 950 patients in at least six participating centers will be included. Consecutive intubated and ventilated adult intensive care patients with an anticipated ventilation duration of minimal 24 hours will be recruited at ICU admission and onset of ventilation.

Methods: Patients will be randomized to receive either: 'routine nebulisation', i.e. nebulisation of mucolytics and bronchodilators, administered every 6 hours (i.e., 4 times per day) for the complete duration of ventilation, or 'nebulisation on strict clinical indications only', i.e. nebulisation of mucolytics in case of occurrence of persistent thick and tenacious sputum, and only after active humidification is set. Nebulisation of bronchodilators in case of occurrence of bronchospasm and only when signs and symptoms of bronchospasm (wheezing, increased airway pressures, increasing airway resistance, up sloping curve of de end tidal CO2 monitoring) are confirmed. The decision to start nebulisation should be evaluated daily. In case the clinical indication no longer exists, the therapy should be stopped.

Patients will be randomly assigned in a 1:1 ratio to one of both nebulisation strategies within 24 hours after ICU admission and intubation, and only if informed consent is signed by the patient or the patient's legal representative. Randomization will be performed using a dedicated, password protected, SSL-encrypted website. Randomization sequence is generated by a dedicated computer randomization software program using random block sizes and is stratified per center. Due to the nature of the intervention blinding of the caregivers is not possible. Data analysis will be performed blinded for the type of intervention.

Standard care: standard care is provided following local guidelines of the participating centers. Recommendations made for mechanical ventilation: Attending physicians are advised to use lung-protective ventilation strategies, including the use of lower tidal volumes (≤ 6 mL/kg predicted body weight) and/or lower airway pressures (≤ 30 cmH2O). Levels of positive end-expiratory pressure (PEEP) and inspired oxygen (FiO2) are titrated on partial pressure of oxygen (PaO2), preferably using a PEEP/ FiO2-table. If spontaneous ventilation is well tolerated it is used from then till the end of ventilation. Thereafter, weaning from ventilation is performed by stepwise lowering of pressure-support level. Daily assessment of the patient's readiness to wean will be performed.

Monitoring: monitoring of patient safety and reviewing of safety issues is performed by a designated independent Data Safety and Monitoring Board (DSMB). The DSMB watches over the ethics of conducting the study in accordance with the Declaration of Helsinki. All (serious) adverse events (SAE) will be collected by the local investigators and sent in to a designated SAE manager, who presents the events to the DSMB for evaluation.

Interim analysis: An interim analysis for safety will be performed after the first one third (193) and two thirds (388) of the study population, respectively, are included and have completed follow up for the primary outcome. The main concern is the occurrence of tube related incidents in the non-nebulized group, development of ventilator associated pneumonia in the nebulisation group. Serious adverse events (SAEs) such as death, ventilator associated pneumonia, ARDS, new onset ventricular tachyarrhythmia with hemodynamic instability wherefore an intervention is indicated or tube occlusion that are possibly related to study intervention will be compared.

Data collection: Data will be collected at inclusion, daily till day 28 after both ICU admission and intubation and at day 90 after both ICU admission and intubation. Data collection will be performed by an investigator blinded for the randomization group, except on day 90 if the patient is discharged. In that case follow-up will be performed by telephone. Data will be coded by a patient identification number (PIN) of which the code will be kept safe at the local sites. The data will be transcribed by local investigators into an internet based electronic case record form (CRF).

Sample size calculation: Group size calculation is focused on demonstrating non-inferiority. When the sample size in each group is 445 (890 patients in total), an one-sided non-inferiority test (targeted at 0.05) for log-transformed normalized data has 80% power to reject the null hypothesis that the number of ventilator-free days (VFDs) in the intervention group (nebulisation on strict clinical indication) is inferior to the number of VFDs in the control group (routine nebulisation) by a margin of 10% and a coefficient of variation of 0.70, in favor of the alternative hypothesis that the number of VFDs in the intervention group is non-inferior. The choice for a margin of 10% is motivated by what we consider acceptable from a clinical point of view as the maximal acceptable reduction of the ventilator-free period for non-inferiority. Clinically this margin means that an increase of > 10% in the duration of mechanical ventilation will reduce the ventilator free days with > 12 hours (calculated over the mean duration of mechanical ventilation of 5 days) which will be considered inferior, assuming that the data will be analyzed in the log scale using t-test for differences in means at the 5% level. To allow for an anticipated drop out of approximately 5%, a number of 475 (950 in total).

As this is a randomized controlled trial, we expect that randomization in this large study population will sufficiently balance the baseline characteristics. However if imbalance occurs, a Cox proportional hazard model will be used and adjusted accordingly.

The effect of nebulisation on the primary outcome will be investigated in pre-specified subgroups based on humidification method (active or passive), different type of nebulisers and continuous versus breath actuated nebulisation.

Time to event variables: Time to event variables of interest (mortality, extubation, tracheotomy, VAP, ARDS, tube occlusion) are analyzed using Cox regression and visualized by Kaplan-Meier.

If the 95% CI upper bound for inferiority of the nebulized-on-indication group is < 10%, the null hypothesis of inferiority is rejected. If the non-inferiority criterion is satisfied, then superiority for the primary endpoint, the number of ventilator free days will be tested.

Organization: The study is conducted by FP, JB, MJS and SMvdH. SMvdH and FP will lead the project. They provide assistance to the participating clinical sites in trial management, record keeping and data management. Local investigators in each site will perform randomization, supervise data collection and ensure adherence to Good Clinical Practice during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year or older
* Expected duration of intubation and ventilation > 24 hours
* Written informed consent

Exclusion Criteria:

* Age less than 18 years
* Ventilation before present ICU admission (though short-term ventilation in the emergency room or in the operation room for general anesthesia during surgery is allowed)
* Suspected or confirmed pregnancy
* Diagnosed with lung diseases for which inhalation therapy and/or oral steroids are used
* Diagnoses of: Guillain-Barré syndrome, complete spinal cord lesion or amyotrophic lateral sclerosis, Multiple Sclerosis, Myasthenia Gravis
* Known allergy for acetylcysteine or salbutamol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2014-07; Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days at day 28 | day 28 after ICU admission and intubation
  The number of ventilator-free days (VFDs) is defined as the number of days from day 1 to day 28 after ICU admission and start of mechanical ventilation on which a patient breathes without assistance of the ventilator if the period of unassisted breathing lasted at least 24 consecutive hours. Patients who die or are mechanically ventilated longer than this period are assigned zero ventilator-free days.

SECONDARY OUTCOMES:
Length of stay | day 28 and day 90 after ICU admission and intubation
  length of stay (ICU and hospital)
Mortality | day 28 and day 90 after ICU admission and intubation
  ICU and hospital mortality
Pulmonary complications | daily until detubation or day 28
  Pulmonary complications will include but are not limited to: incidence of Ventilator-associated Pneumonia (VAP); incidence of secondary acute respiratory distress syndrome (ARDS); atelectasis;
Side effects | daily until detubation or day 28
  Side effects of nebulization of mucolytics and/or bronchodilators (due to nebulization itself, or as a result of exposure to the nebulized agents);

OTHER OUTCOMES:
Health care related costs | until detubation or day 28
  Health care related costs, including costs of ventilation, stay in ICU and/or hospital, cumulative use of sedative drugs and neuromuscular blocking agents, use of tracheostomies, and costs of ventilator-associated pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, Prof Dr MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (7):
- Netherlands (7):
  - Amphia Ziekenhuis Breda, Breda, North Brabant
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Academic Medical Center, Amsterdam, North Holland
  - Isala, Zwolle, Overijssel
  - Sint Antonius Ziekenhuis, Nieuwegein, Utrecht
  - Rijnstate Ziekenhuis, Arnhem
  - MC Haaglanden, The Hague

REFERENCES:
- [Derived] van Meenen DMP, Algera AG, Schuijt MTU, Simonis FD, van der Hoeven SM, Neto AS, Abreu MG, Pelosi P, Paulus F, Schultz MJ; for the NEBULAE; PReVENT; RELAx investigators. Effect of mechanical power on mortality in invasively ventilated ICU patients without the acute respiratory distress syndrome: An analysis of three randomised clinical trials. Eur J Anaesthesiol. 2023 Jan 1;40(1):21-28. doi: 10.1097/EJA.0000000000001778. Epub 2022 Nov 18. PMID 36398740
- [Derived] van der Hoeven S, Ball L, Constantino F, van Meenen DM, Pelosi P, Beenen LF, Schultz MJ, Paulus F; NEBULAE-investigators. Effect of routine vs on-demand nebulization of acetylcysteine with salbutamol on accumulation of airway secretions in endotracheal tubes: substudy of a randomized clinical trial. Intensive Care Med Exp. 2020 Dec 18;8(Suppl 1):71. doi: 10.1186/s40635-020-00351-x. PMID 33336283
- [Derived] van Meenen DMP, van der Hoeven SM, Binnekade JM, de Borgie CAJM, Merkus MP, Bosch FH, Endeman H, Haringman JJ, van der Meer NJM, Moeniralam HS, Slabbekoorn M, Muller MCA, Stilma W, van Silfhout B, Neto AS, Ter Haar HFM, Van Vliet J, Wijnhoven JW, Horn J, Juffermans NP, Pelosi P, Gama de Abreu M, Schultz MJ, Paulus F. Effect of On-Demand vs Routine Nebulization of Acetylcysteine With Salbutamol on Ventilator-Free Days in Intensive Care Unit Patients Receiving Invasive Ventilation: A Randomized Clinical Trial. JAMA. 2018 Mar 13;319(10):993-1001. doi: 10.1001/jama.2018.0949. PMID 29486489
- [Derived] van der Hoeven SM, Binnekade JM, de Borgie CA, Bosch FH, Endeman H, Horn J, Juffermans NP, van der Meer NJ, Merkus MP, Moeniralam HS, van Silfhout B, Slabbekoorn M, Stilma W, Wijnhoven JW, Schultz MJ, Paulus F. Preventive nebulization of mucolytic agents and bronchodilating drugs in invasively ventilated intensive care unit patients (NEBULAE): study protocol for a randomized controlled trial. Trials. 2015 Sep 2;16:389. doi: 10.1186/s13063-015-0865-0. PMID 26329352